CLINICAL TRIAL: NCT04600102
Title: SCANLOAD: The Effect of Limb Loading on Lower Limb Geometry
Status: Withdrawn | Type: Observational
Why Stopped: Study related activities were delayed due to the COVID pandemic and then terminated to focus on higher priority efforts.
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jason Wilken, Principal Investigator, University of Iowa
Other Study IDs: 201907735
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Foot Injuries and Disorders
Keywords: Ankle Foot Orthosis; Adult; 3D Limb Scanning; Limb Geometry; Limb Loading
MeSH Terms: conditions — Foot Injuries; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- GROUP 1: Healthy able-bodied individuals with no history of lower extremity trauma.
  Interventions: Device: Structure Sensor
- GROUP 2: Individuals with unilateral, below knee functional deficits that require an AFO for daily activities (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease).
  Interventions: Device: Structure Sensor

INTERVENTIONS:
Device: Structure Sensor — A 3D representation of each participant's lower limb geometry will be obtained using a Structure Sensor scanner (Occipital, Inc.) which uses an infrared structured light projector to construct a 3D image of an object. The scanner is connected to an iPad; to operate the user rotates the iPad camera around the desired object. In seconds, the entire geometry is digitally reconstructed.

SUMMARY:
Orthotists currently use a range of weight bearing conditions when casting or scanning a patient's limb during the Ankle foot orthosis (AFO) fitting process. This variability in clinical practice is the result of differing opinions regarding the best method for fitting, and a limited understanding of how weight bearing affects the resulting geometry. Few studies have been performed to determine the effect of weight bearing on resulting geometry, or the consistency of the geometry obtained. In this study we seek to evaluate the effect of foot loading on lower limb geometry and the consistency of measurements using low-cost 3D scanning technology, with implications for fitting AFOs.

DETAILED DESCRIPTION:
Two groups of subjects will be recruited for this study. The first group (Group 1) will consist of healthy, able-bodied individuals with no history of lower extremity trauma. The second group (Group 2) will consist of individuals with unilateral, below-knee functional deficits that require an AFO for daily activities (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease).

We will obtain a brief medical history to identify major medical conditions or prior injuries that could influence limb geometry and lead to reliance on an AFO for Group 2 participants.

A 3D representation of each participant's lower limb geometry will be obtained using a Structure Core scanner (Occipital, Inc.), which uses an infrared structured light projector to construct a 3D image of an object. The scanner is connected to an iPad; to operate the scanner, the user rotates the iPad camera around the desired object. In seconds, the entire geometry is digitally reconstructed. Measurements will be evaluated using digital imaging analysis software (Standard Cyborg, Inc.). The different conditions being tested are full weight bearing, partial weight bearing, and non-weight bearing. The effect of limb loading on multiple measures of limb geometry will be evaluated. Limb measurements will include 1) width of the metatarsal heads, 2) width of the calcaneus, 3) foot length, 4) foot height, 5) arch height, 6) medial-lateral width between ankle malleoli, 7) minimum circumference above the ankle malleoli, 8) maximum calf circumference , 9) medial-lateral width of the knee condyles 10) anterior-posterior width at mid patellar tendon, 11) distance from bottom of foot to tibial tubercle.

ELIGIBILITY:
GROUP 1

Patient Inclusion criteria

* Ages: 18-75
* Healthy individuals without a current complaint of lower extremity pain, spine pain, active infections or medical or neuromusculoskeletal disorders that have limited participation in work or exercise in the last 6 months
* Ability to perform a full squat without pain
* Able to read and write in English and provide written informed consent

Patient Exclusion criteria

* Diagnosed moderate or severe brain injury
* Diagnosis of a physical or psychological condition that would preclude testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
* Current complaint of pain or numbness in the spine
* Uncorrected visual or hearing impairments that limit the ability to understand or comply with instructions given during testing
* Require an assistive device
* Open/unhealed wounds on lower extremity.
* Body mass index (BMI) above 35

GROUP 2

Patient Inclusion criteria

* Ages: 18-75
* Daily AFO use to address unilateral below knee functional deficits (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease)
* Ability to stand independently without use of an assistive device (Cane, crutch, etc)
* Ability to safely bear full body weight on affected limb without use of an AFO or other protection
* Able to read and write in English and provide written informed consent

Patient Exclusion criteria

* Use of an AFO that crosses the knee (includes Knee brace or similar)
* Open/unhealed wounds on lower extremity
* Uncorrected visual or hearing impairments that limit the ability to understand or comply with instructions given during testing
* Body mass index (BMI) above 35
* Diagnoses of a moderate to severe brain injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of subjects will be recruited for this study. The first group (Group 1) will consist of healthy, able-bodied individuals with no history of lower extremity trauma. The second group (Group 2) will consist of individuals with unilateral, below-knee functional deficits that require an AFO for daily activities (e.g. fracture, muscle and/or nerve injury, ankle arthritis, or peripheral neurologic disease).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Width of the metatarsal heads | Less than 2 days
  Distance from the medial aspect of the first metatarsal head to the lateral aspect of the fifth metatarsal head.
Width of the calcaneus | Less than 2 days
  Distance from the medial aspect of calcaneus parallel to lateral aspect of calcaneus.
Foot length | Less than 2 days
  Distance from the most posterior aspect of calcaneus to the most anterior toe (1st or 2nd).
Foot height | Less than 2 days
  Distance from the most superior point on the foot distal to the tibialis anterior insertion.
Arch height | Less than 2 days
  Dorsum height at 50% foot length.
Medial-lateral ankle malleoli width | Less than 2 days
  Distance from the lateral malleolus to the medial malleolus.
Minimum ankle circumference | Less than 2 days
  Minimum ankle circumference above the ankle malleoli. Must be less than 10 cm proximal to the ankle malleoli.
Maximum calf circumference | Less than 2 days
  Maximum calf circumference greater that 5 cm distal to the knee condyles.
Width of the knee condyles | Less than 2 days
  Distance from the medial condyle to the lateral condyle.
Anterior-posterior width at patella | Less than 2 days
  Distance from mid patellar tendon to a parallel point most posterior on the back of the knee.
Tibial tubercle height | Less than 2 days
  Distance from the floor to tibial tubercle.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No